CLINICAL TRIAL: NCT05763940
Title: Efficacy of OmegaBoost to Increase Omega-3 Levels Particularly Eicosapentaenoic Acid (EPA) and Docosahexaenoic Acid (DHA) in Healthy Individuals as Compared to the Leading Omega-3 Softgel and the Leading Omega-3 Gummy
Brief Title: Efficacy of OmegaBoost to Increase Omega-3 Levels in Healthy Individuals
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University of Health Sciences (Other)
Collaborators: Guardion Health Sciences, Inc. (Industry)
Responsible Party: Principal Investigator, Pinakin Davey, Principle Investigator, Western University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: GHS.002
Record Dates: First submitted 2023-02-26; First posted 2023-03-10 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Dry Eye Syndromes; Age-Related Macular Degeneration; Omega 3 Index
Keywords: Omega-3s; Docosahexaenoic acid; DHA; Eicosapentaenoic acid; EPA; OmegaBoost; Omega Index test
MeSH Terms: conditions — Dry Eye Syndromes; Macular Degeneration

STUDY DESIGN:
Intervention Model Description: Parallel treatment group participants will be randomly assigned either the experimental interventions;
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OmegaBoost (QD) (Experimental): Participants assigned the study supplement OmegaBoost, taken once daily (QD).
  Interventions: Dietary Supplement: OmegaBoost
- OmegaBoost (BID) (Experimental): Participants assigned the study supplement OmegaBoost, taken twice daily (BID).
  Interventions: Dietary Supplement: OmegaBoost
- Nature Made (soft gel) (Active Comparator): Participants assigned the Nature Made (soft gel), taken twice daily.
  Interventions: Dietary Supplement: Nature Made (soft gel)
- Nature Made (gummy) (Active Comparator): Participants assigned the Nature Made (gummy), taken twice daily.
  Interventions: Dietary Supplement: Nature Made (gummy)

INTERVENTIONS:
Dietary Supplement: OmegaBoost — An ultra-pure omega-3 fish oil supplement with no fishy aftertaste and no fish burps.
  10x more omega-3 from fish oil than the leading omega-3 gummies. Gel bites have better absorption than ordinary, hard-to-swallow fish oil pills.
  Arms: OmegaBoost (BID); OmegaBoost (QD)
Dietary Supplement: Nature Made (soft gel) — A commercially-available omega-3 soft gel formula
  Arms: Nature Made (soft gel)
Dietary Supplement: Nature Made (gummy) — A commercially-available omega-3 formula in gummy form
  Arms: Nature Made (gummy)

SUMMARY:
The purpose of this study is to determine increases in the Omega Index test indicating optimal Omega-3s particularly eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) levels for overall systemic benefits including healthy cardiovascular health and cholesterol levels as shown in the OmegaIndex (OmegaQuant) research.

ELIGIBILITY:
Inclusion Criteria:

* not currently taking Omega-3 supplements or fish oils
* able to swallow softgel or chew gummies nutritional supplement daily for a 12 week period
* able to make four (4) follow-up visits

Exclusion Criteria:

* allergy to fish or seafood
* h/o Atrial fibrillation, or at risk of Afib
* h/o congestive heart failure, heart disease, or prior myocardial infarction and/or cerebrovascular accident
* noncompliance with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2022-05-25 (Actual); Primary Completion 2024-05-25 (Estimated); Study Completion 2024-06-25 (Estimated)

PRIMARY OUTCOMES:
Mean Changes in Omega-3 Index (OmegaQuant) | Baseline, 4 weeks, 8 weeks, and 12 weeks
  OmegaQuant provides Omega Index which is a percentage of omega 3 fatty acids particularly eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in the erythrocytes. The baseline values of OmegaIndex will be compared to repeated measurements obtained at at a 4-, 8- and 12-week. The OmegaQuant labs in Sioux Falls, SD analyze the blood samples to obtain omega-3 levels, omega-6 fatty acids, cis-Monounsaturated Fatty Acids, saturated fatty acids, trans fatty acids. Additionally, arachidonic acid to eicosapentaenoic acid ratio and omega 3 to omega 6 ratios will be calculated
Mean Changes in omega 3 to omega 6 ratios | Baseline, 4 weeks, 8 weeks, and 12 weeks
  The baseline values of omega 3 to omega 6 ratios provided by the blood erythrocyte testing performed the OmegaQuant test will be compared to repeated measurements obtained at a 4-, 8- and 12-week.

SECONDARY OUTCOMES:
Mean Changes in General Health Questionnaire | Baseline, 4 weeks, 8 weeks, and 12 weeks
  Eligible participants will be asked to complete the General Health Questionnaire during each visit to monitor secondary observational improvements and overall compliance. The questionnaire will assess: overall health & wellbeing, overall mood, energy level, stress, mental focus, joint health; along with changes in skin, hair, nails, and dry eye (if applicable). With a lower score considered to be a worse outcome
Mean changes to Hb a1c with Omega Boost supplementation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  For the once daily group Baseline Hba1c is evaluated and will be repeated at various time points that is 4, 8 and 12 weeks. The groups will be compared. A reduction or decrease in values over time is considered an improvement.
Mean changes to total cholesterol with Omega Boost supplementation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  For the once-daily group, baseline total cholesterol is evaluated and will be repeated at various time points that is 4 weeks, 8 weeks, and 12 weeks. The groups will be compared. A reduction or decrease in values over time is considered an improvement.
Mean changes to low-density lipoprotein with Omega Boost supplementation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  For the once-daily group, baseline low-density lipoprotein is evaluated and will be repeated at various time points which are 4 weeks, 8 weeks, and 12 weeks. The groups will be compared. A reduction or decrease in values over time is considered an improvement.
Mean changes to high-density lipoprotein with Omega Boost supplementation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  For the once-daily group baseline high-density lipoprotein is evaluated and will be repeated at various time points that is 4 weeks, 8 weeks, and 12 weeks. The groups will be compared. An increase in values over time is considered an improvement.
Mean changes to triglycerides with Omega Boost supplementation | Baseline, 4 weeks, 8 weeks, and 12 weeks
  For the once-daily group baseline triglycerides is evaluated and will be repeated at various time points which are 4 weeks, 8 week, and 12 weeks. The groups will be compared. A reduction or decrease in values over time is considered an improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Pinakin Gunvant Davey, PhD, OD, Principal Investigator — Western University of Health Sciences
Locations (1):
- Western University of Health Sciences, Pomona, California, United States

IPD SHARING:
Plan to Share IPD: No